CLINICAL TRIAL: NCT03663361
Title: Addressing Neuromuscular Deficits for Improved Outcomes in Ankle Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phillip Gribble (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Phillip Gribble, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 44172; DM170430 (Other Grant/Funding Number: US Army Medical Research Acquisition Activity (USAMRAA))
Record Dates: First submitted 2018-06-14; First posted 2018-09-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Ankle Sprains
Keywords: ankle sprain, sensorimotor, rehabilitation, osteoarthritis
MeSH Terms: conditions — Ankle Injuries; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMART Intervention (Experimental): The SMART intervention will utilize the elements of the Standard of Care intervention, and will also include "Sensorimotor Improvements" and other specific additions that will focus on sensory inputs, motor outputs, and integration of the sensory and motor pathways.
  Interventions: Other: SMART Intervention
- Standard of Care Intervention (Active Comparator): The Standard of Care intervention will include restoration of ankle joint range of motion, strength and functional movement.
  Interventions: Other: Standard of Care Intervention

INTERVENTIONS:
Other: SMART Intervention — Ankle rehabilitation with the addition of sensorimotor components
  Arms: SMART Intervention
Other: Standard of Care Intervention — Ankle rehabilitation focused on restoring range of motion, strength and balance
  Arms: Standard of Care Intervention

SUMMARY:
The purpose of this project is to compare a novel sensorimotor ankle rehabilitation training (SMART) protocol for Lateral ankle sprains (LASs) against a standard of care (SOC) protocol to determine if it is more successful at producing successful one-year outcomes and lower rates of re-injury and improved health. This will address the identified needs for evidence-support and reintegration strategies to improve understanding of the management of patient rehabilitation strategies throughout the rehabilitation process following neuromusculoskeletal injury. The project will validate an innovative rehabilitation approach while providing metrics of success using a variety of clinical and innovative markers.

DETAILED DESCRIPTION:
Background: Ankle injuries are the most common musculoskeletal injuries in the military and civilian populations, creating a substantial time loss that equates to a $5.5 billion annual financial burden. Up to 70% who sustain a lateral ankle sprain (LAS) will develop chronic ankle instability (CAI), with persistent functional disability and injury recurrence. Over 70% of CAI cases will develop early onset post-traumatic ankle joint osteoarthritis (PTOA), with consequent deteriorations in physical activity and health-related quality of life. Given the rate of injuries and discharge rates in the military, the need to deliver improved care to disrupt the path to PTOA is warranted. Our preliminary data demonstrates deficits in central nervous system (CNS) function in patients with CAI, which supports the inclusion of sensorimotor tasks into rehabilitation as an effective means to improve lingering dysfunction and decrease disability in patients with CAI. However, to our knowledge, no investigation has employed these sensorimotor techniques in rehabilitation for acute LAS patients. Therefore, the purpose of this study is to demonstrate the effectiveness of a sensorimotor ankle rehabilitation training (SMART) protocol compared to a standard of care (SOC) protocol at improving clinical and novel outcomes, which will associate with lower rates of LAS re-injury and development of CAI during a 12-month follow-up period. The proposed project is aligned with multiple FY17-18 JPC-8/CRMRP NMSIRRA Focus Areas (i.e. Limited understanding of the management of patient rehabilitation strategies throughout the rehabilitation process following neuromusculoskeletal injury) and Identified Areas of Emphasis (i.e. Develop and evaluate innovative rehabilitation techniques for Service members with neuromusculoskeletal injuries).

Hypotheses: Hypothesis 1.1: Compared to the SOC, LAS patients participating in the SMART program will have improved clinical outcomes at the time of return to full activity. Hypothesis 1.2: Compared to the SOC, LAS patients participating in the SMART program will have improved clinical outcomes and lower LAS re-injury rates at the 6-month follow-up. Hypothesis 1.3: Compared to the SOC, LAS patients participating in the SMART program will have improved clinical outcomes, lower LAS re-injury rates, and less ankle joint cartilage turnover at the 12-month follow-up. Hypothesis 2.1: Compared to the SOC, LAS patients participating in the SMART program will have improved central nervous system function at the time of return to activity, and at the 6-month and 12-month follow-ups. Hypothesis 3.1: Improved mechanistic measures in these innovative outcomes will help explain the success from SMART on the clinical outcomes and ankle joint integrity at the 12-month follow-up.

Specific Aims and Objectives: Our primary purpose is to compare a novel SMART protocol against a SOC protocol to determine if it is more successful at producing successful one-year outcomes and lower rates of re-injury after acute LAS. Specific Aim #1: Determine if SMART improves clinical outcomes (patient-reported function and quality of life, LAS re-injury rates, postural control, ankle ROM) and ankle joint integrity (articular cartilage turnover) in LAS patients. Specific Aim #2: Determine if SMART improves innovative measures of CNS function (corticospinal excitability and brain white matter integrity) in LAS patients. Specific Aim #3: Delineate the association between explanatory mechanistic measures (corticospinal excitability and brain white matter integrity) and the hypothesized improvements in clinical and ankle joint integrity in LAS patients receiving SMART.

Research Strategy: Using a prospective cohort study design, we will compare clinical and CNS outcome measures between cohorts that do or do not develop CAI during the 12 months following an acute LAS from University of Kentucky, University of North Carolina, and Fort Bliss/William Beaumont Army Medical Center. Patients initiating rehabilitation for acute LAS will be randomly assigned to either a SOC or a SMART protocol. Testing will be performed when patients are cleared to return to full duty/activity, and 6 and 12 months after return to duty/activity to determine success in clinical and innovative outcomes.

Military Benefit and Impact: The proposed research study will directly translate to improved clinical outcomes following LAS and prevention of CAI and ankle PTOA. Our work will confirm the need for more comprehensive physical therapy for LAS that addresses sensorimotor deficits that persist commonly after completion of a SOC treatment, bringing a significant clinical impact. This will alleviate financial burdens and time-loss from the common injuries sustained to the ankle, translating into more LAS patients experiencing optimal short-term re-integration and long-term sustained performance, achieving the ultimate goal of "Total Readiness".

ELIGIBILITY:
Inclusion Criteria:

* initiating rehabilitation for a first time acute grade I, II, or III LAS
* have sustained within 72 hours of study enrollment
* diagnosed by a physician, medic, athletic trainer, physical therapist, or other providing medical coverage in operational environments as having sustained a LAS

Exclusion Criteria:

* personal or familial history of epilepsy or seizures
* history of migraine headaches
* ocular foreign body, increased intracranial pressure, open head injury or significant closed head injury
* cochlear implants
* implanted brain stimulators, aneurysm clips or other metal in the head (except mouth)
* implanted medication pumps, pacemakers or intracardiac lines
* current medication with tricyclic anti-depressants, neuroleptic agents or other drugs that lower seizure threshold
* history of diagnosed major psychiatric disorder
* history of illicit drug use
* current alcohol abuse or currently withdrawing from alcohol abuse
* history of heart disease

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Ankle re-injury rate | 12 months
  The number of patient reported re-sprains of the ankle. The outcomes will be assessed at 12 months post-rehabilitation discharge (ie. return to activity).
Change in mental quality of life | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as the sum total from 8 questions. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in physical quality of life | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as the sum total from 8 questions . Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in physical activity | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a score from 0-10, with 10 being the highest level of self-reported physical activity. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in self-reported Functional Ankle Instability | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a score from 0-37 on the Identification of Functional Ankle Instability (IdFAI), with 0 indicating no self-reported ankle instability. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in self-reported Ankle Instability | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a score from 0-5 on the Ankle Instability Instrument (AII), with 0 indicating no self-reported ankle instability. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in self-reported Ankle Disability | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a percentage score from 0-100% on the Foot and Ankle Ability Measure (FAAM), with 100% indicating no self-reported ankle disability. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in dynamic balance | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are reported as linear reach distance normalized to leg length, which are presented as a percentage score, with higher percentage scores representing better dynamic balance. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in ankle dorsiflexion Range of Motion | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a linear distance with larger values representing more estimated joint range of motion. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in corticomotor Excitability - Active Motor Threshold | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented in millivolts with a higher number representing a lower level of cortical excitability. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in corticomotor Excitability - Cortical Silent Period | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a time value in milliseconds with a higher number representing a lower level of cortical excitability. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in Spinal Excitability | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a ratio with a smaller ratio representing a lower level of spinal excitability. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in White Mater Structural Integrity | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a scalar value ranging from 0-1.0 with lower values representing a greater loss of white mater structural integrity. Group means and standard deviations will be reported. TThe outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in Ankle cartilage relaxation | rehabilitation discharge visit, 6 and 12 months post-discharge
  T1rho -magnetic resonance imaging of the superior aspect of the talus in the ankle will be performed. Participant images will be assessed by a blinded observer and scored as a the amount of time required to achieve relaxation. The data are presented in milliseconds. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.
Change in Ankle Articular Cartilage Turnover | rehabilitation discharge visit, 6 and 12 months post-discharge
  Data are presented as a time value in seconds with longer values representing a greater amount of articular cartilage turnover. Group means and standard deviations will be reported. The outcomes will be assessed at the rehabilitation discharge visit and 6 and 12 months post-discharge and reported as change scores over time.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Gribble, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No